CLINICAL TRIAL: NCT00500045
Title: "Retrospective Study of Niacin (as a Vasodilator), Combined With a Topical Steroid (for Macular Edema), For CRVO, HRVO, BRVO."
Brief Title: Retrospective Study of the Effectiveness and Safety of Niacin and Steroid Eye Drops for Retinal Vein Occlusions
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The PI retired/left the institution. Efforts were made to contact the PI but were unsuccessful.
Sponsor: Palo Alto Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAMF 08-51
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Central Retinal Vein Occlusion; Branch Retinal Vein Occlusion
Keywords: CRVO; HRVO; BRVO
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Oral niacin
  Interventions: Drug: nicotinic acid

INTERVENTIONS:
Drug: nicotinic acid — niacin 1500 mg po qd
  Other Names: niacin

SUMMARY:
The aim of this study is to develop a less risky, yet effective and more sustainable treatment for retinal vein occlusions than the current commonly used approach of repeated intravitreal triamcinolone acetonide (Kenalog) injections. The types of retinal vien occlusion that are being studied include central (CVRO), hemi-retinal (HRVO),and branch (BRVO) retinal vein occlusion. Niacin, (Nicotinic Acid, not Nicotinamide) a B-vitamin, has lipid lowering and vasodilating properties. The combination of Niacin and Prednisolone Acetate steroid eye drops as a non-invasive treatment approach was developed by the Principal Investigator. The Niacin dilates the retinal vessels, hopefully encouraging earlier collateral vessel formation aimed at bypassing the venous obstruction, thus restoring venous outflow. The Prednisolone Acetate steroid eye drops are aimed at reducing vascular leakage and therefore the macular edema in the eye while the Niacin is taking effect.

DETAILED DESCRIPTION:
A spontaneous improvement was noted in some patients who were experiencing deteriorating retinal vein occlusions. A chart review and questioning of the patients revealed that the addition of Niacin by the Internist seemed to be the factor that was bringing about the vision improvement.

The Niacin has vasodilating properties, and it is postulated that as the Niacin dilates the retinal vessels, it will encourage earlier collateral vessel formation that will bypass the venous obstruction, and restore venous outflow. The prednisolone steroid eye drops will hopefully reduce the macular edema in the eye.

This is a retrospective study conducted by chart review of up to 45 patients who have undergone treatment with 1500 mg per day of oral Niacin (Nicotinic acid) with or without topical steroid eye drops, Prednisolone acetate (Pred Forte) for the treatment of retinal vein occlusion central (CRVO), hemi-retinal (HRVO), branch (BRVO). The retrospective chart review of patients seen by Dr. Michael Gaynon will go back to 1998 and will continue through the present time. All patients with vision impairment caused by deteriorating retinal vein occlusion, and who were or will be prescribed the Niacin with or without Pred Forte treatment will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have central retinal vein occlusion, hemi-retinal vein occlusion or branch retinal vein occlusion.

Exclusion Criteria:

* Patients with active gout or high levels of uric acid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gaynon, MD, Principal Investigator — Palo Alto Medical Foundation
Locations (1):
- Palo Alto Medical Foundation Department of Ophthalmology, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Oral niacin
  nicotinic acid: niacin 1500 mg po qd
  0 participants started and completed in each arm/group. The PI has retired and left the institution. Efforts were made to contact the PI but were unsuccessful. No study data are available for any results modules.
Period: Overall Study
Arm/Group | Treatment
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 0 participants analyzed for the overall number of baseline participants. The PI has retired and left the institution. Efforts were made to contact the PI but were unsuccessful. No study data are available for any results modules.
Groups:
- Treatment: Oral niacin
  nicotinic acid: niacin 1500 mg po qd
  0 participants analyzed for the overall number of baseline participants. The PI has retired and left the institution. Efforts were made to contact the PI but were unsuccessful. No study data are available for any results modules.
Arm/Group | Treatment
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: An Improvement in Vision in the the Treatment Patients, as Measured by an Increase of 15 Letters on the Early Treatment Diabetic Retinopathy Study (EDTRS) Vision Chart.
Description: 0 participants analyzed for the overall number of participants analyzed. The PI has retired and left the institution. Efforts were made to contact the PI but were unsuccessful. No study data are available for any results modules.
Time Frame: one year
Population: 0 participants analyzed for the overall number of participants analyzed. The PI has retired and left the institution. Efforts were made to contact the PI but were unsuccessful. No study data are available for any results modules.
Groups:
- Treatment: Oral niacin
  nicotinic acid: niacin 1500 mg po qd
  0 participants analyzed for the overall number of participants analyzed. The PI has retired and left the institution. Efforts were made to contact the PI but were unsuccessful. No study data are available for any results modules.
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: A Decrease in the Thickness of the Retina
Description: as for outcome 1
Time Frame: one year
Population: as for outcome 1
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: 0 participants at risk (for each arm/group in both serious and other adverse events). The PI has retired and left the institution. Efforts were made to contact the PI but were unsuccessful. No study data are available for any results modules.
Groups:
- Adverse Events: 0 participants at risk (for each arm/group in both serious and other adverse events). The PI has retired and left the institution. Efforts were made to contact the PI but were unsuccessful. No study data are available for any results modules.
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The PI has retired and left the institution. Efforts were not successful in obtaining data for the study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No